CLINICAL TRIAL: NCT05322967
Title: Chronotherapy in Hypertension - a Study of Blood Pressure Levels Following Intake of Antihypertensive Medication in the Morning or at Bedtime
Brief Title: Effect of Chronotherapy on Blood Pressure - Time of Intake of Blood Pressure Lowering Drugs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Swedish Heart Lung Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: VGFOUREG-939529
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-04

CONDITIONS: Hypertension; Drug Therapy; Primary Health Care
Keywords: Cross-over study
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Participants are randomized in the initial phase to take their ordinary anti-hypertensive medication in the morning or at bedtime for 8 weeks. Then the participants are switching to the alternative intervention during 8 weeks in the second phase of the study.
Who Masked: Outcomes Assessor
Masking Description: It is not possible to mask patients, care provider or investigators but the outcome assessors are masked for allocation of patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning intake (Active Comparator): Intake of antihypertensive medication in the morning
  Interventions: Other: Time of ordinary antihypertensive medication intake
- Bedtime intake (Active Comparator): Intake of antihypertensive medication at bedtime
  Interventions: Other: Time of ordinary antihypertensive medication intake

INTERVENTIONS:
Other: Time of ordinary antihypertensive medication intake — Time of ordinary antihypertensive medication intake

SUMMARY:
A randomized clinical trials with cross-over design to evaluate changes in blood pressure, renal function (creatinine, estimated glomerular filtration), LDL and HDL-cholesterol after taking antihypertensive drugs in the morning or at bedtime. Blood pressure will be estimated by ambulatory blood pressure measurements. There will be a shift in time of drug intake after 8 weeks for each participant. Approximately 100 individuals aged 40-75 years and on stable anti-hypertensive treatment and blood pressure <150/95 mm Hg will be recruited. No new drugs will be introduced during the study.

DETAILED DESCRIPTION:
High blood pressure (hypertension, HT) is very common and can lead to serious cardiovascular complications and premature death. Despite effective drug treatment many patients do not reach the blood pressure goal. No new antihypertensive drugs have been developed lately, so there is a need for other strategies to increase attainment of goals and diminish the rate of complications. The circadian rhythm can affect sleep, body temperature, hormone levels, metabolism and the effect of drugs. The impact of antihypertensive treatment in the short and long run was described in a large randomized study in primary health care where individuals with hypertension were randomly assigned to take the drugs in the morning or at bedtime. Intake at bedtime resulted in lower blood pressure, better kidney function and lower LDL-cholesterol. Further, after a mean time follow-up of 6 years a 50% reduction of cardiovascular death was seen. There was by time running a difference in antihypertensive drugs and also co-morbidity between the groups. Despite this, there is a need to investigate if chronotherapy might play a role in antihypertensive care.

The aim of the study is to investigate the effect of intake of drugs in the morning compared to at bed-time.

Methods: Patients 40-75 years, will be recruited from two primary health care centers and one clinic of internal medicine. Medical history, current medication will be recorded. Office blood pressure, body height and weight, ECG and ambulatory blood pressure measurement (ABPM) will be performed. Blood will be analyzed for fasting blood glucose, LDL and HDL-cholesterol and creatinine.

After inclusion in the study the patients are randomly, by clinic, allocated to take their antihypertensive drugs in the morning or at bed-time during 8 week. The ordinary medication is used during the study period. The patients are instructed to keep a diary on wake-up and bed-times, side effects, sleep quality and other experiences during therapy. After 8 weeks the investigations at base-line are repeated and a visual analogue scale on sleep, daytime tiredness and urine voiding is recorded. The patients shift to intake of medication on the opposite time of day for 8 weeks. The study is completed with a repeated investigation as above. The analyses of data is performed by researchers of the team that are not aware of the patients' allocation. The diaries will be a base for later in-depth-interviews with a part of the patients. The analyses will be intention-to-treat using appropriate methods for the data. Office blood pressure, blood lipids and kidney function at baseline, 8 and 16 weeks, as well as sleep duration, urine voiding at night will be analyzed. ABPM will be analyzed using mean blood pressure around-the-clock, daytime and nighttime blood pressure, dipping and morning surge.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertension
* Stable antihypertensive treatment at least 8 weeks prior to inclusion
* One to four antihypertensive drugs

Exclusion Criteria:

* Atrial fibrillation/flutter
* Diabetes
* Previous stroke or TIA
* Heart failure
* Ischemic heart disease
* Peripheral artery disease
* Malignant disease with less than one year expected survival
* Inability to follow study protocol (for instance shift work)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-25 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
24 hours blood pressure changes between 8 and 16 weeks. | 8 and 16 weeks
  Ambulatory blood pressure changes between 8 and 16 weeks. Systolic and diastolic mean blood pressure level.
Change of dipping of blood pressure between 8 and 16 weeks. | 8 and 16 weeks
  Ratio between daytime and nighttime blood pressure registered after 8 and 16 weeks. Systolic and diastolic mean blood pressure level.

SECONDARY OUTCOMES:
Daytime blood pressure changes between 8 and 16 weeks. | 8 and 16 weeks
  Ambulatory daytime blood pressure registered after 8 and 16 weeks. Systolic and diastolic mean blood pressure level.
Nighttime blood pressure changes between 8 and 16 weeks. | 8 and 16 weeks
  Ambulatory nighttime blood pressure registered after 8 and 16 weeks. Systolic and diastolic mean blood pressure level.
Office blood pressure changes between 8 and 16 weeks. | 8 and 16 weeks
  Office blood pressure registered after 8 and 16 weeks. Systolic and diastolic mean blood pressure level.
Difference in morning surge of blood pressure between 8 and 16 weeks. | 8 and 16 weeks
  Occurrence of morning (yes/no)
Difference in LDL cholesterol levels between 8 and 16 weeks. | 8 and 16 weeks
  LDL cholesterol changes according to time of intake of antihypertensive drugs
Difference in HDL cholesterol levels between 8 and 16 weeks. | 8 and 16 weeks
  HDL cholesterol changes according to time of intake of antihypertensive drugs
Difference in total cholesterol levels between 8 and 16 weeks. | 8 and 16 weeks
  Total cholesterol changes according to time of intake of antihypertensive drugs
Difference in p-creatinine levels between 8 and 16 weeks. | 8 and 16 weeks
  P-creatinine changes according to time of intake of antihypertensive drugs

OTHER OUTCOMES:
Difference in score of Epworth sleepiness scale between 8 and 16 weeks | 8 and 16 weeks
  Epworth sleepiness scale score registered by the patients according to time of antihypertensive drug intake
Perceived side effects 8 weeks | 8 weeks
  Perceived side effects registered by the patients (VAS) according to time of antihypertensive drug intake
Perceived side effects 16 weeks | 16 weeks
  Perceived side effects registered by the patients (VAS) according to time of antihypertensive drug intake

CONTACTS AND LOCATIONS:
Overall Officials: Karin Manhem, Prof, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (3):
- Sweden (3):
  - Sahlgrenska University Hospital, Mölndal, Gothenburg
  - Närhälsan Billingen Primary Health Care Centre, Skövde
  - Närhälsan Norrmalm Primary Health Care Centre, Skövde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hermida RC, Crespo JJ, Dominguez-Sardina M, Otero A, Moya A, Rios MT, Sineiro E, Castineira MC, Callejas PA, Pousa L, Salgado JL, Duran C, Sanchez JJ, Fernandez JR, Mojon A, Ayala DE; Hygia Project Investigators. Bedtime hypertension treatment improves cardiovascular risk reduction: the Hygia Chronotherapy Trial. Eur Heart J. 2020 Dec 21;41(48):4565-4576. doi: 10.1093/eurheartj/ehz754. PMID 31641769
- [Background] Hermida RC. Sleep-time ambulatory blood pressure as a prognostic marker of vascular and other risks and therapeutic target for prevention by hypertension chronotherapy: Rationale and design of the Hygia Project. Chronobiol Int. 2016;33(7):906-36. doi: 10.1080/07420528.2016.1181078. Epub 2016 May 24. PMID 27221952
- [Background] Fujiwara T, Hoshide S, Yano Y, Kanegae H, Kario K. Comparison of morning vs bedtime administration of the combination of valsartan/amlodipine on nocturnal brachial and central blood pressure in patients with hypertension. J Clin Hypertens (Greenwich). 2017 Dec;19(12):1319-1326. doi: 10.1111/jch.13128. Epub 2017 Nov 5. PMID 29106031
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Bilo G, Grillo A, Guida V, Parati G. Morning blood pressure surge: pathophysiology, clinical relevance and therapeutic aspects. Integr Blood Press Control. 2018 May 24;11:47-56. doi: 10.2147/IBPC.S130277. eCollection 2018. PMID 29872338
- [Background] Bowles NP, Thosar SS, Herzig MX, Shea SA. Chronotherapy for Hypertension. Curr Hypertens Rep. 2018 Sep 28;20(11):97. doi: 10.1007/s11906-018-0897-4. PMID 30267334
- [Background] Callaway E, Ledford H. Medicine Nobel awarded for work on circadian clocks. Nature. 2017 Oct 2;550(7674):18. doi: 10.1038/nature.2017.22736. No abstract available. PMID 28980662
- [Background] 2018 Practice Guidelines for the management of arterial hypertension of the European Society of Hypertension and the European Society of Cardiology: ESH/ESC Task Force for the Management of Arterial Hypertension: Erratum. J Hypertens. 2019 Feb;37(2):456. doi: 10.1097/HJH.0000000000002026. No abstract available. PMID 30640882